CLINICAL TRIAL: NCT04062825
Title: Interaction of HIV/Platelets and HIV-platelets/Lymphocytes in HIV Patients Under cART Treatment But Immunological Non Responders
Brief Title: Interaction Between HIV and Platelets
Acronym: PLAQUEVIH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 19CCN-VIH-Plaquettes
Record Dates: First submitted 2019-07-01; First posted 2019-08-20 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: HIV Seropositivity
Keywords: HIV; platelets; lymphocytes; cART; InRs
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- VIH positive patients without lymphoma: 200 VIH positive patients without lymphoma
- VIH positive patients with lymphoma: 20 VIH positive patients with lymphoma
- healthy volunteers: 20 healthy volunteers

SUMMARY:
The investigators propose that the lack of immune response in InR is driven by HIV-containing platelets that might interact with macrophages and CD4+ T-cells although by different mechanisms. In the one hand, HIV-sheltering platelets might fuel tissue HIV macrophage and in turn T cell reservoirs as observed in InRs and/or maintain a low-level viral replication in macrophages, sustaining a persistent inflammatory profile on in these cells. In the other hand,HIV-sheltering platelets might induce CD4+ T-cells dysfunctions via platelets/ectosomes, although without promoting platelet-to-T-cell HIV transfer/infection, thereby increasing the number of peripheral inflammatory TH17 cells and a TH17/Treg unbalance as observed in InRs.

Main Objectives:

i) To characterize and the molecular and functional level the platelet factors implicated in HIV transfer to tissue-like macrophages as well as in the immunomodulatory activity of HIV-containing platelets on macrophages and CD4+ T-cells.

ii) To interrogate the transfer of HIV-containing platelet-derived mRNA and microRNA to tissue-like macrophages and CD4+ T-cells as one major mechanism of target cell immunomodulation.

iii) To investigate the therapeutic potential of anti-platelet aggregation/activation agents (e.g. Abciximab), known to block platelet-immune cell interaction, in improving immune cell functions in vitro and promoting immunological recovery in vivo.

DETAILED DESCRIPTION:
The investigators have recently shown that infectious HIV is carried by platelets in the blood of HIV-infected patients which failed to respond immunologically to cART despite viral suppression (Immunological nonresponders, InRs) and that platelets can mediate HIV transmission to macrophages in vitro, in line with our recent description of HIV reservoir occurrence and establishment in macrophages in cART-suppressed patients. Around 20% of the overall cART-treated patients are InRs that fail to reconstitute their competent immune status despite treatment observance with prolonged viral suppression. The causes of this immunological failure remain unclear and no treatment is available to improve the health of InRs, which are at higher risk of AIDS and non-AIDS morbidity and mortality. The poor immunological recovery in InRs is mainly driven by a sustained low CD4+ T-cell counts that relies on persistent inflammation and immune activation affecting T-cell population profile.

Platelets are cleared by tissue macrophages in vivo in physiological or inflammatory contexts, what could represent a route for HIV to establish reservoirs in macrophages. We have shown that HIV sheltered in platelets can transfer infection to macrophages, in a process blocked by anti-αIIb/ β3 antibody Abciximab. This infection is productive as in turn, infection spreads replication-competent virus to non-infected CD4+ T-cells. This viral spread may increase the blood T-cell HIV reservoir, a hallmark of immunological failure as observed in InRs. In contrast, HIV-containing platelets fail to directly infect CD4+ T, unless infection is forced by the fusion inducer polybrene. Thus, in contrast to macrophages, CD4+ T cells are not targeted by HIV enclosed in platelets.

However, HIV-containing platelets might immunomodulate CD4+ T cell functions thereby triggering the immunological failure observed in cART-suppressed patients. Hence, platelet-T-cell conjugates form in the blood of HIV patients, suggesting that HIV-containing platelets could downregulate T-cell functions. Platelets are known to express adhesive proteins that not only promote platelet aggregation responsible for primary hemostasis, but also to mediate interactions with leukocytes, driving either inhibition of proliferation and differentiation of CD4+ T-cells into TH17, crucial in mediating chronic inflammation. Platelets can also shed microvesicles (ectosomes) which directly contact these lymphocytes, driving TH17 polarization of CD4+ T-cells and in turn an unbalanced TReg/TH17 ratio characteristic of InRs. Such TReg/TH17 unbalance might reflect a persistent inflammatory state that could translate in a cytotoxic/antiproliferative effect on CD4+ T-cells and ultimately immunological failure.

Very recently, we found that the number of platelets-CD4+ T-cells conjugates circulating in the blood of cART-treated HIV-infected patients is increased in InRs (virally suppressed and <350 CD4+T-cells/μl) compared with immunological responders (IR, >500 CD4+T-cells/μl). In addition, conjugates form more with TH17 in InR compared with IR, whereas conjugates form equally with TReg in the two InR and IR patients groups. These results indicate that InRs not only present a strong probability to have HIV-containing platelets but are also prone to form platelets-TH17 cells conjugates, suggesting a causal connection between association of HIV with platelets and platelet-driven immunomodulation of CD4+T-cells toward a TH17 profile. Whether these platelet-TH17 conjugates we observed form with full platelets or platelet ectosome (that both harbor CD41 used as platelet marker in our conjugate analyses) remains unknown.

Importantly, HIV RNA is only detected in circulating CD4+ T-cell reservoirs when latent proviral DNA is reactivated, suggesting that platelet-containing HIV does not conjugate with CD4+T cell in InR patients but rather with bystander platelets or platelet ectosomes (lacking HIV). Thus, immunomodulation of CD4+T cells in InRs might result from the interaction with these bystander platelet/ectosomes or ectosomes shed from HIV-containing platelets.

Platelets have been shown to exchange mRNA upon interaction with immune cells and tumors . Furthermore, transfer of functional mRNA and microRNA is so far demonstrated to be mediated by platelet ectosomes, targeting macrophage/monocytic and epithelial cells. Thus, transfer of messenger RNAs or microRNAs from platelets/ectosomes to macrophages and/or CD4+ T-cells could be the mechanism of platelet-dependent immunomodulation of target leukocytes. Platelets display a repertoire of mainly pro-inflammatory microRNAs such as miRNA-155 and miRNA-326, involved in NF-κB-mediated inflammatory macrophage responses 25 and TH17 cell-polarization. These miRNAs could be differentially expressed in platelets containing HIV and their eventual transfer to target immune cells could participate in immune cell dysfunction as observed in InRs. Furthermore, αIIb/ β3 mRNA are platelet-specific transcripts conserved in circulating platelets throughout their life-span, and can be exploited to tag leukocytes targeted by mRNA/microRNA of HIV-containing platelets.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* aged ⩾ 18 years;
* patients who can read and understand information document.

For VIH positive patients without lymphoma:

* VIH positive patients with negative or positive viral load under cART since 1 year;
* patient under cART.

For VIH positive patients with lymphoma:

* VIH positive patient with negative viral load under cART since 1 year;
* patient with lymphoma.

For Healthy Volunteers:

* VIH negative patient (control) already included in clinical trial;
* patient major without haematological pathology.

Exclusion Criteria:

* patient < 18 years;
* Unable to read and understand information document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 VIH positive patients without lymphome + 20 VIH positive patients with lymphome + 20 healthy volunteers (VIH negative).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
CD4 number will be determined | at 48 month
  Immunological response status based on the presence-absence of HIV in platelets during follow-up: CD4 number will be determined by flow cytometry.
VIH level in platelet will be quantified | at 48 month
  Immunological response status based on the presence-absence of HIV in platelets during follow-up: VIH level in platelet will be quantified by flow fich and PCR.

SECONDARY OUTCOMES:
potential interaction between platelets and lymphocytes | 12-36 months
  in vitro characterization of interaction between lymphocytes and platelets by microscopy. The cells will be stained with specific antibodies
potential interaction between platelets and lymphocytes | 12-36 months
  in vitro characterization of interaction between lymphocytes and platelets by flow cytometry. The cells will be stained with specific antibodies
analyze if the interaction can be blocked by anti GPIIbIIIa | 12-36 months
  anti GPIIbIIIa will be added in culture dish with platelets and lymphocytes. Analysis of inhibition of interaction will be performed by flow cytometry.
analyze if the interaction can be blocked by anti GPIIbIIIa | 12-36 months
  anti GPIIbIIIa will be added in culture dish with platelets and lymphocytes. Analysis of inhibition of interaction will be performed by microscopy.
HIV expression on bone marrow smear | 1-48 months
  cells from bone marrow will be spread on a slide; and presence of HIV will be performed with an anti HIV anti body
soluble factors secretion | 12-36 months
  HIV+ platelets will be cultivated with donor's CD4 lymphocytes of. By ELISA and/or Bioplex, the secretion of soluble factors (cytokines, chemokines, soluble receptors), secreted by Lymphocytes in the culture medium will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Capron, MD, Principal Investigator — Service Hématologie Immunologie, Hôpital Ambroise Paré; MORGANE BOMSEL, MD, Study Director — Unité CNRS UMR 8104, INSERM U1016, Laboratoire Entrée muqueuse du VIH et Immunité muqueuse, Département Infection, Immunité et Inflammation, Institut Cochin Université Paris Descartes
Locations (1):
- Service Hématologie Immunologie, Hôpital Ambroise Paré, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganor Y, Real F, Sennepin A, Dutertre CA, Prevedel L, Xu L, Tudor D, Charmeteau B, Couedel-Courteille A, Marion S, Zenak AR, Jourdain JP, Zhou Z, Schmitt A, Capron C, Eugenin EA, Cheynier R, Revol M, Cristofari S, Hosmalin A, Bomsel M. HIV-1 reservoirs in urethral macrophages of patients under suppressive antiretroviral therapy. Nat Microbiol. 2019 Apr;4(4):633-644. doi: 10.1038/s41564-018-0335-z. Epub 2019 Feb 4. PMID 30718846
- [Background] Real F, Sennepin A, Ganor Y, Schmitt A, Bomsel M. Live Imaging of HIV-1 Transfer across T Cell Virological Synapse to Epithelial Cells that Promotes Stromal Macrophage Infection. Cell Rep. 2018 May 8;23(6):1794-1805. doi: 10.1016/j.celrep.2018.04.028. PMID 29742434
- [Background] Kaufmann GR, Perrin L, Pantaleo G, Opravil M, Furrer H, Telenti A, Hirschel B, Ledergerber B, Vernazza P, Bernasconi E, Rickenbach M, Egger M, Battegay M; Swiss HIV Cohort Study Group. CD4 T-lymphocyte recovery in individuals with advanced HIV-1 infection receiving potent antiretroviral therapy for 4 years: the Swiss HIV Cohort Study. Arch Intern Med. 2003 Oct 13;163(18):2187-95. doi: 10.1001/archinte.163.18.2187. PMID 14557216
- [Background] Baker JV, Peng G, Rapkin J, Krason D, Reilly C, Cavert WP, Abrams DI, MacArthur RD, Henry K, Neaton JD; Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). Poor initial CD4+ recovery with antiretroviral therapy prolongs immune depletion and increases risk for AIDS and non-AIDS diseases. J Acquir Immune Defic Syndr. 2008 Aug 15;48(5):541-6. doi: 10.1097/QAI.0b013e31817bebb3. PMID 18645520
- [Background] Kelley CF, Kitchen CM, Hunt PW, Rodriguez B, Hecht FM, Kitahata M, Crane HM, Willig J, Mugavero M, Saag M, Martin JN, Deeks SG. Incomplete peripheral CD4+ cell count restoration in HIV-infected patients receiving long-term antiretroviral treatment. Clin Infect Dis. 2009 Mar 15;48(6):787-94. doi: 10.1086/597093. PMID 19193107
- [Background] Chene G, Sterne JA, May M, Costagliola D, Ledergerber B, Phillips AN, Dabis F, Lundgren J, D'Arminio Monforte A, de Wolf F, Hogg R, Reiss P, Justice A, Leport C, Staszewski S, Gill J, Fatkenheuer G, Egger ME; Antiretroviral Therapy Cohort Collaboration. Prognostic importance of initial response in HIV-1 infected patients starting potent antiretroviral therapy: analysis of prospective studies. Lancet. 2003 Aug 30;362(9385):679-86. doi: 10.1016/s0140-6736(03)14229-8. PMID 12957089
- [Background] Deeks SG, Kitchen CM, Liu L, Guo H, Gascon R, Narvaez AB, Hunt P, Martin JN, Kahn JO, Levy J, McGrath MS, Hecht FM. Immune activation set point during early HIV infection predicts subsequent CD4+ T-cell changes independent of viral load. Blood. 2004 Aug 15;104(4):942-7. doi: 10.1182/blood-2003-09-3333. Epub 2004 Apr 29. PMID 15117761
- [Background] Hunt PW, Martin JN, Sinclair E, Bredt B, Hagos E, Lampiris H, Deeks SG. T cell activation is associated with lower CD4+ T cell gains in human immunodeficiency virus-infected patients with sustained viral suppression during antiretroviral therapy. J Infect Dis. 2003 May 15;187(10):1534-43. doi: 10.1086/374786. Epub 2003 Apr 23. PMID 12721933
- [Background] Marziali M, De Santis W, Carello R, Leti W, Esposito A, Isgro A, Fimiani C, Sirianni MC, Mezzaroma I, Aiuti F. T-cell homeostasis alteration in HIV-1 infected subjects with low CD4 T-cell count despite undetectable virus load during HAART. AIDS. 2006 Oct 24;20(16):2033-41. doi: 10.1097/01.aids.0000247588.69438.fd. PMID 17053349
- [Background] Nunes-Alves C, Nobrega C, Behar SM, Correia-Neves M. Tolerance has its limits: how the thymus copes with infection. Trends Immunol. 2013 Oct;34(10):502-10. doi: 10.1016/j.it.2013.06.004. Epub 2013 Jul 16. PMID 23871487
- [Background] Wilson EM, Singh A, Hullsiek KH, Gibson D, Henry WK, Lichtenstein K, Onen NF, Kojic E, Patel P, Brooks JT, Sereti I, Baker JV; Study to Understand the Natural History of HIV/AIDS in the Era of Effective Therapy (SUN Study) Investigators. Monocyte-activation phenotypes are associated with biomarkers of inflammation and coagulation in chronic HIV infection. J Infect Dis. 2014 Nov 1;210(9):1396-406. doi: 10.1093/infdis/jiu275. Epub 2014 May 9. PMID 24813472
- [Background] Ballem PJ, Belzberg A, Devine DV, Lyster D, Spruston B, Chambers H, Doubroff P, Mikulash K. Kinetic studies of the mechanism of thrombocytopenia in patients with human immunodeficiency virus infection. N Engl J Med. 1992 Dec 17;327(25):1779-84. doi: 10.1056/NEJM199212173272503. PMID 1435932
- [Background] Grozovsky R, Hoffmeister KM, Falet H. Novel clearance mechanisms of platelets. Curr Opin Hematol. 2010 Nov;17(6):585-9. doi: 10.1097/MOH.0b013e32833e7561. PMID 20729731
- [Background] Hatano H, Hayes TL, Dahl V, Sinclair E, Lee TH, Hoh R, Lampiris H, Hunt PW, Palmer S, McCune JM, Martin JN, Busch MP, Shacklett BL, Deeks SG. A randomized, controlled trial of raltegravir intensification in antiretroviral-treated, HIV-infected patients with a suboptimal CD4+ T cell response. J Infect Dis. 2011 Apr 1;203(7):960-8. doi: 10.1093/infdis/jiq138. PMID 21402547
- [Background] Green SA, Smith M, Hasley RB, Stephany D, Harned A, Nagashima K, Abdullah S, Pittaluga S, Imamichi T, Qin J, Rupert A, Ober A, Lane HC, Catalfamo M. Activated platelet-T-cell conjugates in peripheral blood of patients with HIV infection: coupling coagulation/inflammation and T cells. AIDS. 2015 Jul 17;29(11):1297-308. doi: 10.1097/QAD.0000000000000701. PMID 26002800
- [Background] Starossom SC, Veremeyko T, Yung AW, Dukhinova M, Au C, Lau AY, Weiner HL, Ponomarev ED. Platelets Play Differential Role During the Initiation and Progression of Autoimmune Neuroinflammation. Circ Res. 2015 Oct 9;117(9):779-92. doi: 10.1161/CIRCRESAHA.115.306847. Epub 2015 Aug 20. PMID 26294656
- [Background] Miossec P, Kolls JK. Targeting IL-17 and TH17 cells in chronic inflammation. Nat Rev Drug Discov. 2012 Oct;11(10):763-76. doi: 10.1038/nrd3794. PMID 23023676
- [Background] Rodriguez-Munoz A, Martinez-Hernandez R, Ramos-Levi AM, Serrano-Somavilla A, Gonzalez-Amaro R, Sanchez-Madrid F, de la Fuente H, Marazuela M. Circulating Microvesicles Regulate Treg and Th17 Differentiation in Human Autoimmune Thyroid Disorders. J Clin Endocrinol Metab. 2015 Dec;100(12):E1531-9. doi: 10.1210/jc.2015-3146. Epub 2015 Oct 19. PMID 26480286
- [Background] De Benedetto I, Masetti M, Fabbiani M, Biasin M, Muscatello A, Squillace N, Clerici M, Trabattoni D, Gori A, Bandera A. Higher Levels of Peripheral Th17 T CD4+ Cells Are Associated With Immunological Non Response in HIV-Infected Patients Under Effective ART. J Acquir Immune Defic Syndr. 2018 Apr 15;77(5):e45-e47. doi: 10.1097/QAI.0000000000001627. No abstract available. PMID 29315114
- [Background] Deeks SG. HIV infection, inflammation, immunosenescence, and aging. Annu Rev Med. 2011;62:141-55. doi: 10.1146/annurev-med-042909-093756. PMID 21090961
- [Background] Joosse SA, Pantel K. Tumor-Educated Platelets as Liquid Biopsy in Cancer Patients. Cancer Cell. 2015 Nov 9;28(5):552-554. doi: 10.1016/j.ccell.2015.10.007. PMID 26555171
- [Background] Laffont B, Corduan A, Ple H, Duchez AC, Cloutier N, Boilard E, Provost P. Activated platelets can deliver mRNA regulatory Ago2*microRNA complexes to endothelial cells via microparticles. Blood. 2013 Jul 11;122(2):253-61. doi: 10.1182/blood-2013-03-492801. Epub 2013 May 7. PMID 23652806
- [Background] Risitano A, Beaulieu LM, Vitseva O, Freedman JE. Platelets and platelet-like particles mediate intercellular RNA transfer. Blood. 2012 Jun 28;119(26):6288-95. doi: 10.1182/blood-2011-12-396440. Epub 2012 May 17. PMID 22596260
- [Background] Mann M, Mehta A, Zhao JL, Lee K, Marinov GK, Garcia-Flores Y, Lu LF, Rudensky AY, Baltimore D. An NF-kappaB-microRNA regulatory network tunes macrophage inflammatory responses. Nat Commun. 2017 Oct 11;8(1):851. doi: 10.1038/s41467-017-00972-z. PMID 29021573
- [Background] Rowley JW, Chappaz S, Corduan A, Chong MM, Campbell R, Khoury A, Manne BK, Wurtzel JG, Michael JV, Goldfinger LE, Mumaw MM, Nieman MT, Kile BT, Provost P, Weyrich AS. Dicer1-mediated miRNA processing shapes the mRNA profile and function of murine platelets. Blood. 2016 Apr 7;127(14):1743-51. doi: 10.1182/blood-2015-07-661371. Epub 2016 Jan 14. PMID 26773046
- [Background] Du C, Liu C, Kang J, Zhao G, Ye Z, Huang S, Li Z, Wu Z, Pei G. MicroRNA miR-326 regulates TH-17 differentiation and is associated with the pathogenesis of multiple sclerosis. Nat Immunol. 2009 Dec;10(12):1252-9. doi: 10.1038/ni.1798. Epub 2009 Oct 18. PMID 19838199
- [Background] Ple H, Landry P, Benham A, Coarfa C, Gunaratne PH, Provost P. The repertoire and features of human platelet microRNAs. PLoS One. 2012;7(12):e50746. doi: 10.1371/journal.pone.0050746. Epub 2012 Dec 4. PMID 23226537
- [Background] Podshivalova K, Salomon DR. MicroRNA regulation of T-lymphocyte immunity: modulation of molecular networks responsible for T-cell activation, differentiation, and development. Crit Rev Immunol. 2013;33(5):435-76. doi: 10.1615/critrevimmunol.2013006858. PMID 24099302
- [Background] Fink L, Holschermann H, Kwapiszewska G, Muyal JP, Lengemann B, Bohle RM, Santoso S. Characterization of platelet-specific mRNA by real-time PCR after laser-assisted microdissection. Thromb Haemost. 2003 Oct;90(4):749-56. doi: 10.1160/TH03-02-0095. PMID 14515198
- [Background] Zhu A, Real F, Zhu J, Greffe S, de Truchis P, Rouveix E, Bomsel M, Capron C. HIV-Sheltering Platelets From Immunological Non-Responders Induce a Dysfunctional Glycolytic CD4+ T-Cell Profile. Front Immunol. 2022 Feb 11;12:781923. doi: 10.3389/fimmu.2021.781923. eCollection 2021. PMID 35222352
- [Background] Real F, Capron C, Sennepin A, Arrigucci R, Zhu A, Sannier G, Zheng J, Xu L, Masse JM, Greffe S, Cazabat M, Donoso M, Delobel P, Izopet J, Eugenin E, Gennaro ML, Rouveix E, Cramer Borde E, Bomsel M. Platelets from HIV-infected individuals on antiretroviral drug therapy with poor CD4+ T cell recovery can harbor replication-competent HIV despite viral suppression. Sci Transl Med. 2020 Mar 18;12(535):eaat6263. doi: 10.1126/scitranslmed.aat6263. PMID 32188724